CLINICAL TRIAL: NCT06750484
Title: Open-label Single-arm Phase 2 Trial of Trastuzumab Deruxtecan in Previously Treated HER2-Immunohistochemistry (IHC) 0 Advanced Breast Cancer
Brief Title: Trial of Trastuzumab Deruxtecan in Previously Treated HER2
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Yale University (Other)
Collaborators: Daiichi Sankyo (Industry); AstraZeneca (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2000035049
Record Dates: First submitted 2024-12-16; First posted 2024-12-27 (Actual); Last update posted 2025-10-21 (Actual); Status verified 2025-10

CONDITIONS: Breast Cancer Metastatic
Keywords: HER2-IHC 0
MeSH Terms: interventions — trastuzumab deruxtecan

STUDY DESIGN:
Intervention Model Description: All people enrolled in the study will receive the same treatment and no one will receive a placebo or alternate treatment.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (1):
- Trastuzumab Deruxtecan (Experimental): T-DXd will be administered intravenously every 3 weeks at a dose of 5.4 mg per kilogram of body weight until disease progression, limiting toxicity, withdrawal of consent, or death. For T-DXd, each cycle of treatment will be 21 days. The number of treatment cycles with T-DXd is not fixed.
  Interventions: Drug: Trastuzumab Deruxtecan

INTERVENTIONS:
Drug: Trastuzumab Deruxtecan — Participants will receive the study drug trastuzumab deruxtecan (T-DXd) by IV infusion every 21 days. The number of treatment cycles will depend on how participants respond to treatment.

SUMMARY:
The purpose of this study is to test the good and bad effects of a drug called trastuzumab deruxtecan (T-DXd) in adult patients with metastatic HER2-negative breast cancer and which patients might benefit the most from T-DXd.

DETAILED DESCRIPTION:
HER2 (human epidermal growth factor receptor 2) is a gene that can play a role in the development of breast cancer. Genes like HER2 and the proteins they make influence how a breast cancer behaves and how it might respond to a specific treatment.

A score of 0 on the HER2 immunohistochemistry (IHC) test indicates that breast tissue is HER2-negative. Drugs that fight cancer by targeting the growth of HER2 genes, such as the monoclonal antibody trastuzumab, have not traditionally been used in patients with HER2-negative tumors because trastuzumab works by attaching to HER2 and stopping cancer cells from growing and dividing. However, about half of breast cancers that are categorized as HER2-negative like yours, actually have low expression of HER2. and recent research has shown that newer generations of antibody-drug conjugates like trastuzumab show considerable survival benefit even in tumors that are not classified as HER2-positive.

An antibody-drug conjugates is a combination of a monoclonal antibody like trastuzumab with an anticancer agent like deruxtecan. This combination that interrupts DNA replication in cancer cells. Antibody-drug conjugates like (T-DXd) are designed to target and kill cancer cells while sparing healthy cells.

Prior research that has shown that the antibody-drug conjugate trastuzumab deruxtecan (T-DXd) has outstanding activity and survival benefit in HER2-low breast cancers.

The purpose of this study is to help us learn more about which patients might benefit most from T-DXd through a single-arm, open-label, phase 2 study to assess the safety and efficacy of T-DXd in HER2-negative subjects with unresectable and/or metastatic breast cancer.

The researchers will measure the response to the T-DXd (the percentage of patients with complete response, partial response, stable disease, and progressive disease). Researchers will also look for biomarkers to determine the most accurate way to predict which patients without HER2-positive breast cancer will benefit the most from T-DXd.

T-DXd has been FDA approved to treat adults with unresectable or metastatic HER2-low breast cancer who have received a prior chemotherapy in the metastatic setting or developed disease recurrence during or within six months of completing adjuvant chemotherapy.

Each treatment cycle is 21 days.

ELIGIBILITY:
Inclusion Criteria:

1. Must be competent and able to comprehend, sign, and date an Institutional Review Board (IRB) approved ICF before performance of any study-specific procedures or tests.
2. Men or women ≥18 years old.
3. Pathologically documented breast cancer that is unresectable or metastatic.
4. 4.Tumor biopsies have always shown HER2-IHC 0 (<10% membrane staining, including 0 null and 0 ultralow) in all prior biopsies and never previously HER2-positive (IHC 3+ or ISH+) or HER2-low (1+, or 2+ ISH-) on prior pathology testing according to American Society of Clinical Oncology College of American Pathologists (ASCO-CAP) guidelines.
5. Either HR-positive or HR-negative status of the tumor per ASCO-CAP guidelines are allowed.
6. Patients with HR-positive disease must have progressed or be intolerant to CDK 4/6 inhibitors plus endocrine therapy, and patients with HR-negative disease must have received 1 line of therapy in the metastatic setting (progression on or within 6 months of neoadjuvant or adjuvant therapy will be accounted for as 1 line of prior therapy). There is no limit on number of subsequent lines of therapy for study entry. .
7. Patients must have never been previously treated with any anti-HER2 therapy, including prior trastuzumab deruxtecan, other HER2-directed ADCs, HER2 antibodies or HER2 tyrosine kinase inhibitors
8. Clinical or radiologic progression (during or after most recent treatment) or intolerance to therapy prior to enrollment in this trial
9. Adequate archival tumor sample <3 years-old available for assessment of HER2 status by IHC and by HS-HER2 quantitative assay. If archival tissue is not available or inadequate for assessment (e.g. decalcified bone, cytology, or other), a newly obtained biopsy from a metastatic site (or breast tissue if locally advanced/unresectable disease as the only site of advanced disease) is required on enrolment.
10. Presence of at least 1 measurable lesion based on Response Evaluation Criteria in Solid Tumors (RECIST) version 1.1.
11. ECOG PS ≤ 2.
12. Left ventricular ejection fraction (LVEF) ≥50% within 28 days prior to C1D1.
13. Adequate bone marrow function (Table 1) within 28 days before C1D1, defined as:

    1. Platelet count >≥100,000/mm3 (Platelet transfusion is not allowed within 1 week prior to Screening assessment).
    2. Hemoglobin level ≥9.0 g/dL (red blood cell transfusion is not allowed within 1 week prior to Screening assessment).
    3. Absolute neutrophil count ≥1500/mm3 (granulocyte colony-stimulating factor administration is not allowed within 1 week prior to Screening assessment).
14. Adequate renal function (Table 1) within 28 days before C1D1, defined as:

    a. Creatinine clearance ≥30 mL/min, as calculated using the Cockcroft-Gault Equation.
15. Adequate hepatic function (Table 1) within 28 days before C1D1, defined as:

    1. Aspartate aminotransferase (AST)/alanine aminotransferase (ALT) ≤ 3×ULN (< 5×ULN in participants with liver metastases).
    2. Total bilirubin ≤1.5 × ULN if no liver metastases or <3 × ULN in the presence of documented Gilbert's syndrome (unconjugated hyperbilirubinemia) or liver metastases at baseline.
16. Adequate blood clotting function( defined below) within 28 days before C1D1, defined as International normalized ratio or Prothrombin time and either partial thromboplastin or activated partial thromboplastin time ≤ 1.5 × ULN.

    1. Platelet function greater than or equal to 100000/mm3 (Platelet transfusion is not allowed within 1 week prior to C1D1).
    2. Hemoglobin greater than or equal to 9.0 g/dL NOTE: Participants requiring ongoing transfusions or growth factor support to maintain haemoglobin ≥9.0 g/dL are not eligible. Red blood cell transfusion is not allowed within 1 week prior to C1D1.
    3. Absolute neutrophil count greater than or equal to 1500/mm3. (granulocyte-colony stimulating factor administration is not allowed within 1 week prior to C1D1).
    4. Alanine aminotransferase and aspartate aminotransferase less than or equal to 3×ULN (< 5×ULN in participants with liver metastases).
    5. Total bilirubin less than or equal to 1.5×ULN if no liver metastases or < 3×ULN in the presence of documented Gilbert's syndrome (unconjugated hyperbilirubinemia) or liver metastases at baseline.
    6. Serum albumin greater than or equal to 2.5 g/dL
    7. Creatine clearance greater than or equal to 30 mL/min as determined by Cockcroft Gault (using actual body weight).
    8. International normalised ratio or Prothrombin time and either partial thromboplastin or activated partial thromboplastin time less than or equal to 1.5 x upper limit of normal
17. Adequate treatment washout period before C1D1, defined below:

    1. Major surgery minimum washout period of greater than or equal to 4 weeks
    2. Radiation therapy including palliative stereotactic radiation therapy to chest minimum washout period greater than or equal to 4 weeks
    3. Palliative stereotactic radiation therapy to other anatomic areas including whole brain radiation minimum wash out period of greater than or equal 2 weeks
    4. Anti-Cancer chemotherapy [Immunotherapy (non-antibody based therapy)], hormonal therapy, antibody-based therapy, or retinoid therapy minimum washout period greater than or equal to 3 weeks
    5. Anti-Cancer chemotherapy [Immunotherapy (non-antibody based therapy)], hormonal therapy, antibody-based therapy, or retinoid therapy minimum washout period greater than or equal 3 weeks
    6. Targeted agents and small molecules minimum washout period greater than or equal 2 weeks or 5 half-lives, whichever is longer
    7. Cell-free and Concentrated Ascites Reinfusion Therapy (CART), peritoneal shunt or drainage of pleural effusion, ascites or pericardial effusion minimum washout period greater than or equal to 2 weeks prior to screening assessment
    8. Any monoclonal antibody treatment minimum washout period greater than or equal to 3 elimination half-lives of the inhibitor/antibody
18. Evidence of post-menopausal status or negative serum pregnancy test for females of childbearing potential who are sexually active with a non-sterilized male partner. For women of childbearing potential, a negative result for serum pregnancy test (test must have a sensitivity of at least 25 mIU/mL) must be available at the screening visit and urine beta-human chorionic gonadotropin (β-HCG) pregnancy test prior to each administration of T-DXd. Women of childbearing potential are defined as those who are not surgically sterile (i.e. underwent bilateral salpingectomy, bilateral oophorectomy, or complete hysterectomy) or post-menopausal. Women will be considered post-menopausal if they have been amenorrheic for 12 months without an alternative medical cause.
19. Female patients of childbearing potential who are sexually active with a non-sterilized male partner must use at least one highly effective method of contraception, presented in Table 3 from the time of screening (those using hormonal methods must have been stable on their chosen form of contraception for 3 months prior to study entry) and must agree to continue using such precautions for 7 months after the last dose of T-DXd. Not all methods of contraception are highly effective. Female patients must refrain from breastfeeding while on study and for 7 months after the last dose of T-DXd. Complete heterosexual abstinence for the duration of the study and drug washout period is an acceptable contraceptive method if it is line with the patient's usual lifestyle (consideration must be made to the duration of the clinical trial); however, periodic or occasional abstinence, the rhythm method, and the withdrawal method are not acceptable.
20. Non-sterilized male patients who are sexually active with a female partner of childbearing potential must use a condom from screening to 4 months after the final dose of T-DXd. Complete heterosexual abstinence for the duration of the study and drug washout period is an acceptable contraceptive method if it is in line with the patient's usual lifestyle (consideration must be made to the duration of the clinical trial); however, periodic or occasional abstinence, the rhythm method, and the withdrawal method are not acceptable. It is strongly recommended for the female partners of a male patient to also use at least one highly effective method of contraception throughout this period, as described in Table 3. In addition, male patients should refrain from fathering a child or freezing or donating sperm from the time of enrolment, throughout the study and for 4 months after the last dose of T-DXd. Preservation of sperm should be considered prior to enrolment in this study.
21. Female subjects must not donate, or retrieve for their own use, ova from the time of enrolment and throughout the study treatment period, and for at least 7 months after the final study drug administration. They should refrain from breastfeeding throughout this time. Preservation of ova may be considered prior to enrolment in this study.

Exclusion Criteria:

1. Uncontrolled or significant cardiovascular disease, including any of the following:

   1. History of myocardial infarction within 6 months before enrolment.
   2. History of symptomatic congestive heart failure (New York Heart Association Class II to IV).
   3. Corrected QT interval (QTc) Fridericia prolongation to >470 ms (females) or >450 ms (male) based on average of Screening 12 lead ECG.
2. Uncontrolled or significant respiratory disease criteria, including any of the following:

   1. Has a history of (noninfectious) ILD/pneumonitis that required steroids, has current ILD/pneumonitis, or where suspected ILD/pneumonitis cannot be ruled out by imaging at Screening.
   2. Lung-specific intercurrent clinically significant illnesses including, but not limited to, any underlying pulmonary disorder (e.g. severe asthma, severe chronic obstructive pulmonary disorder, restrictive lung disease, symptomatic, recurrent and uncontrolled pleural effusion etc.)
   3. Any autoimmune, connective tissue or inflammatory disorders, including Rheumatoid arthritis, Sjogren's, and sarcoidosis, where there is documented, or a suspicion of pulmonary involvement at the time of screening. Full details of the disorder should be recorded in the eCRF for participants who are included in the study.
   4. Prior pneumonectomy (complete)
3. Has spinal cord compression or clinically active central nervous system metastases, defined as untreated and symptomatic, or requiring therapy with corticosteroids to control associated symptoms.

   1. Subjects with clinically inactive brain metastases may be included in the study.
   2. Subjects with treated brain metastases that are no longer symptomatic and who require no treatment with corticosteroids may be included in the study if they have recovered from the acute toxic effect of radiotherapy. A minimum of 2 weeks must have elapsed between the end of whole brain radiotherapy and study enrolment.
4. Has history of another primary malignancy, except for:

   1. Malignancy treated with curative intent and with no known active disease ≥5 years before the first dose of IP and of low potential risk for recurrence.
   2. Adequately treated non-melanoma skin cancer or lentigo maligna without evidence of disease.
   3. Adequately treated carcinoma in situ without evidence of disease.
5. Has a history of severe hypersensitivity reactions to either the drug substances or inactive ingredients in the drug product, or history of severe hypersensitivity reactions to monoclonal antibodies.
6. Has an uncontrolled infection requiring ongoing IV antibiotics, IV antivirals, or IV antifungals.
7. Has known history of human immunodeficiency virus (HIV) infection with detectable viral load or CD4 count < 200 cells per cubic millimeter or active hepatitis B ( HBsAg positive) or C (HCV positive RNA) infection.
8. Substance abuse, medical conditions such as clinically significant cardiac or pulmonary diseases or psychological, social, familial, or geographical conditions, that would, in the opinion of the Investigators, increase the safety risk to the subject or interfere with the subject's participation in the clinical study or evaluation of the clinical study results.
9. Has unresolved toxicities from previous anticancer therapy, defined as toxicities (other than alopecia) not yet resolved to Grade ≤1 or baseline. Subjects with chronic Grade 2 toxicities may be eligible per the discretion of the Investigator [e.g., Grade 2 chemotherapy-induced neuropathy, fatigue, residual endocrinopathies from use of immunotherapy such as hypothyroidism/hyperthyroidism, type 1 diabetes, hyperglycemia, adrenal insufficiency, adrenalitis, skin hypopigmentation (vitiligo)].
10. Is pregnant or breastfeeding, or planning to become pregnant.
11. Receipt of live, attenuated vaccine (mRNA and replication deficient adenoviral vaccines are not considered attenuated live vaccines) within 30 days prior to the first exposure to study intervention. Note: Participants, if enrolled, should not receive live vaccine during the study and up to 30 days after the last dose of study intervention.
12. Otherwise considered inappropriate for the study by the Investigator.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2025-06-20 (Actual); Primary Completion 2028-12-31 (Estimated); Study Completion 2028-12-31 (Estimated)

PRIMARY OUTCOMES:
Objective Response Rate | After cycle 3, approximately 63 days
  The confirmed Objective Response Rate to Trastuzumab Deruxtecan by RECIST (Response Evaluation Criteria In Solid Tumors) defined as the cumulative rate of complete response (CR) rate and partial response (PR) rates, evaluated according to mRECIST v1.1

SECONDARY OUTCOMES:
Objective Response Rate (ORR) Comparison by HER2 Status | through study completion, an average of 1 year
  To assess and compare the Objective Response Rates (ORRs) between two subgroups of patients defined by their HER2 status. Patients will be classified into two subgroups: HER2 detectable and HER2 non-detectable. The ORR will be measured based on the proportion of patients in each subgroup who achieve a predefined response (complete response or partial response) to the treatment regimen, according to RECIST (Response Evaluation Criteria in Solid Tumors) criteria.
Correlation between HER2 protein expression | Last follow up visit (40 days [+7] from last dose)
  To explore and evaluate the association between HER2 protein expression value measured by the HS-HER2 assay in the CLIA lab setting with objeective response and clinical benefit from T-DXd.
Progression Free Survival (PFS) | From the date of enrolment to the earliest date of the first objective documentation of radiographic disease progression according to mRECIST version 1.1 or death due to any cause. up to 3 years
  Progression Free Survival based on investigator assessment, in all subjects
Overall Survival (OS) | (every 3 months +/-14 days) for up to 3 years
  Overall Survival in all subjects

CONTACTS AND LOCATIONS:
Overall Officials: Adriana Kahn, M.D., Principal Investigator — Yale University
Locations (1):
- Yale University, New Haven, Connecticut, United States

IPD SHARING:
Plan to Share IPD: No